CLINICAL TRIAL: NCT03802149
Title: Cervical Preparation Using Ulipristal Acetate for Second Trimester Surgical Abortion
Brief Title: Ulipristal Acetate for Cervical Preparation
Acronym: U-Prep
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-48756
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Termination of Pregnancy
Keywords: Ulipristal Acetate; Abortion; Cervical Preparation; Dilation and Evacuation
MeSH Terms: conditions — Dilatation, Pathologic | interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ulipristal Acetate (Experimental): Participants will be administered a one time dose of 90mg ulipristal acetate 18-24-hours prior to dilation and evacuation (surgical abortion) for cervical preparation.
  Interventions: Drug: Ulipristal Acetate

INTERVENTIONS:
Drug: Ulipristal Acetate — 90mg Ulipristal Acetate 18-24-hours prior to dilation and evacuation

SUMMARY:
This is a prospective cohort study exploring a broadened use of ulipristal acetate as a cervical preparation agent for second trimester surgical abortion. Specifically, this pilot study will test the feasibility of using ulipristal as a pharmacologic cervical preparation with adjunct misoprostol prior to surgical abortion.

DETAILED DESCRIPTION:
Second trimester abortion comprises <10% of all induced abortions in the United States but there is still an important need to provide this service to women. Prior to dilation and evacuation (D&E), adequate preparation of the uterine cervix is an important part of preventing complications of the procedure. Commonly, this is done using osmotic dilators that are placed into the uterine cervix but cervical preparation can also be achieved using medications alone. Mifepristone is commonly used for this purpose but its use is regulated and often restricted due to the REMS (Risk Evaluation and Mitigation Strategy) program. The objective of this pilot study is to test the feasibility of using ulipristal, an oral medication similar to Mifepristone, as a medical form of cervical preparation prior to surgical abortion.This is a prospective cohort study investigating the use of ulipristal acetate (UPA) for pharmacologic cervical preparation with adjunct misoprostol prior to second trimester surgical abortion among women who are 16 to 18 6/7 weeks gestational age. Due the mechanism of action of UPA as a selective progesterone receptor modulator (SPRM) being similar to that of mifepristone, a medication known to be effective for cervical preparation, the investigators seek to describe the use of another SPRM for this same purpose. The investigators will conduct a pilot study assessing the feasibility of using UPA for cervical priming and report descriptive measures of its use. Per clinic protocols, patients over 16-weeks gestation attend a consult and cervical preparation appointment the day prior to their procedure. Eligible patients will be offered enrollment. Subjects will receive UPA 90mg one day prior to their procedure and no osmotic dilators. All subjects will receive pre-procedure misoprostol (600mcg 90 minutes prior to procedure). The investigators will observe patients through their planned procedure and report descriptive measures of its use.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 years or older
* Singleton, viable intrauterine pregnancy between 16 to 18 6/7 weeks of gestation (by ultrasound dating performed prior to or same day of enrollment visit)
* Consented for an induced, elective abortion
* English-speaking
* Able to consent for research project
* Willingness to comply with study procedures

Exclusion Criteria:

* Inability to give informed consent
* Contraindications to surgical abortion under moderate sedation
* Allergy or previous unacceptable side effect from study medications
* Multiple gestation
* Intrauterine fetal demise or spontaneous abortion
* Rupture of membranes
* Current cervical insufficiency
* History of liver disease
* Taken a CYP3A4 inhibitor within 5 elimination half-lives of the drug from the procedure
* Pre-dosing abnormal liver function tests
* Patients at increased risk of hepatitis based on a history of any of the following:
* Any history of underlying liver disorder, including hepatitis
* A family history of hepatitis or currently living with a person who has been given a diagnosis of hepatitis
* A history of or currently working as a sex worker
* A history of or currently using IV drugs
* A self-reported history of alcoholic dependency or abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Adequacy of cervical dilation | Intraoperative
  Ease of dilation, measured by visual analog score (0-100mm, 0 being "very easy" and 100 being "very difficult"

SECONDARY OUTCOMES:
Need for additional mechanical dilation | Intraoperative: start of dilation to completion of dilation
  Number of dilator increments in French required to dilate the internal os
Total procedure time | Intraoperative: from speculum placement to speculum removal
  Minutes
Total operative time | Intraoperative: insertion of the first instrument to removal of the last instrument from the uterus
  Minutes
Complications | Intraoperative and postoperative through 8-weeks
  Number of cervical lacerations, uterine perforation, hemorrhage and need for transfer to high level of care
Overall Pain Experienced | 20-minutes postoperative
  0-100mm on visual analog scale
Number of procedures completed as scheduled | Time from enrollment to completion of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Will assess IPD sharing upon request.

REFERENCES:
- [Derived] Peterson SF, Lerma K, Shaw KA, Blumenthal PD. Cervical Preparation Using Ulipristal Acetate With Adjunct Misoprostol in Second-Trimester Surgical Abortions. Obstet Gynecol. 2022 May 1;139(5):907-909. doi: 10.1097/AOG.0000000000004754. Epub 2022 Apr 5. No abstract available. PMID 35576349